CLINICAL TRIAL: NCT03648307
Title: Long-term Effect of Splenectomy on Metabolism, a Retrospective Cohort Study
Brief Title: Long Term Effect of Splenectomy on Metabolism
Status: Completed | Type: Observational
Sponsor: Imam Hossein General Hospital (Other)
Responsible Party: Principal Investigator, Parnian Jabbari, Researcher at Imam Hossein General Hospital, Medical Doctor, Imam Hossein General Hospital
Other Study IDs: ImamHGH
Record Dates: First submitted 2018-08-18; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Trauma Splenic
Keywords: Splenectomy; metabolism; diabetes; stem cells; trauma surgery
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection; Body Mass Index; Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples for lipid profile and Hb A1C
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma splenectomized: Patients who had gone through trauma splenectomy. BMI, lipid profile, blood pressure and glucose tolerance of patients were assessed. Hb A1C and lipid profile were assessed through blood sampling.
  Interventions: Diagnostic Test: Blood sample
- Bowel resection: Patients who had gone through bowel resection due to obstruction. BMI, lipid profile, blood pressure and glucose tolerance of patients were assessed. Hb A1C and lipid profile were assessed through blood sampling.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample for Hb A1C and lipid profile, blood pressure and BMI
  Other Names: BMI and blood pressure measurement

SUMMARY:
Metabolic status of patients who had gone through trauma splenectomy between July 2008 and July 2013 were compared to patients who had gone through bowel resection due to obstruction in the same period of time. all patients were followed up for 5-10 years.

DETAILED DESCRIPTION:
A list was made of patients who had gone through trauma splenectomy or bowel resection due to bowel obstruction in our center between July 2008 and July 2013. Patients were divided into two groups: trauma splenectomy (exposed group) and bowel resection (unexposed group).

All patients were followed up for 5-10 years. Of the 243 splenectomized patients, 90 patients who met our study criteria were willing to participate. Of 152 patients with bowel resection, 64 were willing to participate. Records of patients at the time of surgery were retrieved from hospital archive of patients' records. Patients were invited to an office meeting for assessment of blood pressure, BMI and a general physical examination and history taking. An appointment was made for drawing blood samples for measurement of lipid profile, Hb A1C and fasting blood sugar.

Exclusion criteria:

1. Disturbed lipid profile at the time of surgery, 2. Disturbed blood glucose levels at the time of surgery, 3. History of high blood pressure prior to surgery, 4. Use of any hyperglycemogenic agent during the follow up period, 5. BMI>= 25 at the time of surgery, 6. History of diseases potentially affecting blood glucose, e.g. hyperthyroidism, Cushing syndrome, 7. Accidental pancreatic damage during surgery, 8. Resection of >10 cm of small bowel and 9. History of malignancy or radiotherapy (criteria 8 and 9 were specific to unexposed group).

ELIGIBILITY:
Inclusion Criteria:

* trauma splenectomy or bowel resection due to obstruction between July 2008 and July 2013

Exclusion Criteria:

* disturbed lipid profile at the time of surgery
* disturbed blood glucose at the time of surgery
* history of high blood pressure at the time of surgery
* use of any hyperglcemogenic agent during the follow up
* BMI>= 25 at the time of surgery
* history of diseases that can affect blood glucose levels
* accidental pancreatic damage during surgery
* resection of > 10 cm of small bowel (for bowel resection group)
* history of malignancy or radiotherapy (for bowel resection group)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had gone through bowel resection due to obstruction or trauma splenectomy in Imam Hosein General Hospital between July 2008 and July 2013
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | July 2008- July 2013
  Glucose tolerance was assessed by measuring the Hb A1C of the patients in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Behzad Nemati Honar, professor, Study Director — Imam Hosein General Hospital; Sahar Saeedi, MD, Principal Investigator — Imam Hosein General Hospital

IPD SHARING:
Plan to Share IPD: No
Details of patients identities and data obtained from measurements will not be shared with other researchers.

DOCUMENTS (1):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03648307/Prot_000.pdf